CLINICAL TRIAL: NCT03935893
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Adoptive Transfer of Autologous Tumor Infiltrating Lymphocytes in Patients With Advanced Solid Cancers
Brief Title: Adoptive Transfer of Tumor Infiltrating Lymphocytes for Advanced Solid Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Udai Kammula (Other)
Responsible Party: Sponsor-Investigator, Udai Kammula, Director, Solid Tumor Cell Therapy Program, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-004
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; Colorectal Cancer; Pancreatic Cancer; Sarcoma; Mesothelioma; Neuroendocrine Tumors; Squamous Cell Cancer; Merkel Cell Carcinoma; Mismatch Repair Deficiency; Microsatellite Instability
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Sarcoma; Mesothelioma; Neuroendocrine Tumors; Neoplasms, Squamous Cell; Carcinoma, Merkel Cell; Turcot syndrome; Microsatellite Instability | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: This study will follow the Bayesian basket design proposed by Simon et al (2016). Treatment will be considered active in a specific histology cohort if the response rate is over 20% (phi = 0.2) and not active if the response rate is less than 5% (plo = 0.05).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tumor Infiltrating Lymphocytes (TIL) (Experimental): Patients with locally advanced, recurrent, or metastatic gastric/esophagogastric, colorectal, pancreatic, sarcoma, mesothelioma, neuroendocrine, cutaneous/anal squamous cell, Merkel cell, cancers refractory to systemic therapy, and those with deficient mismatch repair and/or microsatellite instability cancers will receive the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide, followed by infusion of up to 2x10^11 lymphocytes infused through a central vein catheter and administered at a dose of 600,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to a maximum of 6 doses.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL); Drug: Fludarabine + Cyclophosphamide combination

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — TIL are to be infused intravenously through a central vein catheter over 20-30 minutes followed by Aldesleukin, administered at a dose of 600,000 IU/kg (based on total body weight) as an intravenous bolus over a 15-minute period approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to a maximum of 6 doses.
Drug: Fludarabine + Cyclophosphamide combination — Preparative lymphocyte depleting (immunosuppressive) combination regimen consisting of fludarabine and cyclophosphamide administered prior to TIL infusion.
  Other Names: Fludara; Cytoxan

SUMMARY:
This is a Phase 2 study to evaluate the efficacy of a non-myeloablative lymphodepleting preparative regimen followed by infusion of autologous TIL and high-dose aldesleukin in patients with locally advanced, recurrent, or metastatic cancer associated with one of the following cancer types: 1.) gastric/esophagogastric, 2.) colorectal, 3.) pancreatic, 4.) sarcoma, 5.) mesothelioma, 6.) neuroendocrine, 7.) squamous cell cancer, 8.) Merkle cell, 9.) mismatch repair deficient and/or microsatellite unstable cancers, and 10.) patients who have exhausted conventional systemic therapy options by using the objective response rate (ORR).

DETAILED DESCRIPTION:
This Phase 2 study will be conducted in conjunction with companion protocol (Cell Harvest and Preparation to Support Adoptive Cell Therapy Clinical Protocols and Pre-Clinical Studies) as described below:

Cell Preparation:

Patients with evaluable locally advanced, recurrent, or metastatic gastric/esophagogastric, colorectal, pancreatic, sarcoma, mesothelioma, neuroendocrine, cutaneous/anal squamous cell, Merkel cell, cancers refractory to systemic therapy, and those with deficient mismatch repair and/or microsatellite instability cancers who have lesions that can be resected or biopsied with minimum morbidity will undergo resection or biopsy of tumor. TIL will be obtained while enrolled on the companion protocol HCC 17-220 (Cell Harvest and Preparation to Support Adoptive Cell Therapy Clinical Protocols and Pre-Clinical Studies). Separate tumor procurements may be performed under HCC 17-220 protocol to obtain TIL if initial tumor procurements could not successfully generate TIL. The TIL will be grown and expanded for this trial according to standard operating procedures submitted in the IND. The TIL will be assessed for potency by interferon-gamma release.

Treatment Phase:

Once cells exceed the potency requirement and are projected to exceed the minimum number specified in the COA, the patient will be registered on this study and receive the lymphocyte depleting preparative regimen consisting of fludarabine and cyclophosphamide, followed by infusion of up to 2x10^11 lymphocytes (minimum of 1x10^9 cells) and administration of high-dose intravenous aldesleukin. It is anticipated that TIL that meet the COA will not be achievable in approximately 20% of patients who undergo resection. These patients may undergo a second resection to grow TIL, if another suitable lesion exists. Approximately 6 weeks (+/- 2 weeks) after TIL administration, patients will undergo a complete tumor evaluation and evaluation of toxicity and immunologic parameters. Patients will receive one course of treatment. The start date of the course will be the start date of the chemotherapy; the end date will be the day of the first post-treatment evaluation. Patients may undergo a second treatment. Patients will receive no other experimental agents while on this protocol.

ELIGIBILITY:
Inclusion Criteria:

Measurable locally advanced, recurrent, or metastatic cancer associated with one of the following cancer types: 1.) gastric/esophagogastric, 2.) colorectal, 3.) pancreatic, 4.) sarcoma, 5.) mesothelioma, 6.) neuroendocrine, 7.) squamous cell cancer, 8.) Merkle cell, 9.) mismatch repair deficient and/or microsatellite unstable cancers, and 10.) patients who have exhausted conventional systemic therapy options

Patients with locally advanced disease should be unresectable by conventional surgical approaches.

Patients with distant metastatic spread must have previously received approved first-line systemic therapies if they are eligible to receive these treatments.

Patients must be co-enrolled on the companion protocol HCC 17-220 (Cell Harvest and Preparation to Support Adoptive Cell Therapy Clinical Protocols and Pre-Clinical Studies) and have available TIL cultures for therapy.

Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.

Greater than or equal to 18 years of age and less than or equal to age 75

Able to understand and sign the Informed Consent Document

Clinical performance status of ECOG 0 or 1

Life expectancy of greater than three months

Patients of both genders who are of child-bearing potential must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the treatment.

Serology:

* Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen
* Seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.

Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.

Hematology

* Absolute neutrophil count greater than 1000/mm3 without the support of filgrastim
* WBC ≥ 3000/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin > 8.0 g/dl

Chemistry

* Serum ALT/AST ≤ to 3.5 times the upper limit of normal Serum creatinine ≤ to 1.6 mg/dl
* Total bilirubin ≤ to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a clinically manageable level (except for toxicities such as alopecia or vitiligo). (Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less)

Exclusion Criteria:

Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.

Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).

Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).

Active systemic infections (e.g.: requiring anti-infective treatment),

Clinically significant coagulation disorder

Active major medical illnesses deemed clinically significant by the treating physician

History of clinically significant major organ autoimmune disease

Patients with a history of hypothyroidism are eligible

Concurrent systemic steroid therapy.

History of severe immediate hypersensitivity reaction to any of the agents used in this study.

History of active coronary or ischemic symptoms.

Documented LVEF of less than or equal to 45%; note: testing is required in patients with:

* Age > 65 years' old
* Clinically significant atrial and or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second- or third-degree heart block or have a history of ischemic heart disease, chest pain.

Documented FEV1 less than or equal to 60% predicted tested in patients with:

* A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
* Symptoms of respiratory dysfunction

Patients who are receiving any other investigational agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2037-06-30 (Estimated); Study Completion 2038-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Number of patients with Complete Response (CR) + Number of patients with Partial Response (PR) / total number of patients (# with CR + # with PR + # with SD + # with PD), per RECIST v1.1: CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: ≥ 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Progressive Disease (PD): ≥ 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance ≥1 new lesion(s) is considered progression.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | 24 months
  Proportion of patients with complete response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1): Number of patients with Complete Response (CR) / total number of patients (# with CR + # with PR + # with SD + # with PD). CR: disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Progressive Disease (PD): ≥ 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance ≥1 new lesion(s) is considered progression.
Duration of response (DOR) | 24 months
  Time between the initial response to treatment per Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and subsequent disease progression among patients achieving Complete Response (CR) or Partial Response (PR). Per RECIST v1.1, Complete Response (CR): disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Disease control rate (DCR) | 24 months
  Number of patients with Complete Response (CR) + Number of patients with Partial Response (PR) + Number of patients with Stable Disease (SD) / total number of patients (# with CR + # with PR + # with SD + # with PD), per RECIST v1.1. (CR):disappearance of all target lesions.Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Progression-free survival (PFS) | 24 months
  The length of time after TIL infusion treatment that a patient lives with disease that does not progress per RECIST v1.1. Per RECIST, Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall survival (OS) | 24 months
  The length of time from the start of treatment that patients are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Udai S Kammula, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No